CLINICAL TRIAL: NCT06757868
Title: The Effect of Amobarbital on Myocardial Protection and Prognosis in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Amobarbital and Cardiopulmonary Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Doctor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMOC
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cardiopulmonary Bypass
MeSH Terms: interventions — Amobarbital; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amo group (Experimental): amobarbital 1mg/kg is given prior to cardiopulmonary bypass
  Interventions: Drug: Amobarbital
- Mida group (Active Comparator): midazolam 0.1mg/kg is given prior to cardiopulmonary bypass
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Amobarbital — Amobarbital 1mg/kg is given prior to cardiopulmonary bypass
  Other Names: AMO
  Arms: Amo group
Drug: Midazolam — midazolam 0.1mg/kg is given prior to cardiopulmonary bypass
  Other Names: MIDA
  Arms: Mida group

SUMMARY:
Explore the effects of amobarbital on myocardial protection and prognosis in patients undergoing cardiac surgery with cardiopulmonary bypass, investigate the new usage of old drugs, and provide reliable clinical scientific basis for its potential value in better clinical treatment.

DETAILED DESCRIPTION:
AMO is a short acting complex I blocker that blocks mitochondrial complex I between flavoprotein and ubiquitin, and its blocking effect can be rapidly reversed. Our study is to explore the effects of amobarbital on myocardial protection and prognosis in patients undergoing cardiac surgery with cardiopulmonary bypass, investigate the new usage of old drugs, and provide reliable clinical scientific basis for its potential value in better clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-65 years old, undergo elective cardiac surgery with extracorporeal circulation.
* ASA II-III;
* surgical duration is 3-6 hours;
* Sign the informed consent form

Exclusion Criteria:

* BMI less than 18 kg/m2 or greater than 30 kg/m2;
* Individuals with a history or potential history of drug abuse or alcohol dependence;
* Preoperative use of sedatives or analgesics;
* Individuals with severe liver and kidney dysfunction;
* Individuals who are allergic or potentially allergic to barbiturates;
* Patients with coagulation dysfunction, endocrine disorders, or other conditions that affect hemodynamic status;
* Participated in other clinical studies in the past 3 months;
* The researchers believe that participants who are not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac recurrence time | 1 hour after heart beat recurrence
  Stop extracorporeal circulation until heart beat time

SECONDARY OUTCOMES:
extubation time | 1day
  time from stopping anesthetics to extubation
cTnI | 2 days
  Using enzyme-linked immunosorbent assay (ELISA) to detect serum cardiac troponin I (cTnI) in patients

CONTACTS AND LOCATIONS:
Overall Officials: Aihua Du, Dr, Study Chair — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No